CLINICAL TRIAL: NCT03104959
Title: Use of N-acetyl Cysteine (NAC) in Alleviation or Prevention of Hangover Symptoms; Independent Alcohol Consumption Protocol
Brief Title: Use of NAC in Prevention of Hangover Symptoms; Independent Alcohol Consumption Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to enroll sufficient number of participants
Sponsor: St. Luke's Hospital and Health Network, Pennsylvania (Other)
Responsible Party: Principal Investigator, Holly Stankewicz, D.O., attending physician and faculty emergency medicine residency, St. Luke's Hospital and Health Network, Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SLUHN2015-105
Record Dates: First submitted 2016-12-12; First posted 2017-04-07 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Prevention of Hangover Using N-Acety Cysteine
Keywords: hangovers; N-acetyl cysteine; alcohol
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Healthy volunteers consume alcohol independently and estimate number of drinks then apply Vick's vapor rub under nose and take placebo capsules based on number of drinks consumed and fill out a Hangover Symptom Scale the next morning
  Interventions: Other: placebo
- N-acetyl cysteine (Experimental): Healthy volunteers consume alcohol independently and estimate number of drinks then apply Vick's vapor rub under nose and take N-Acetyl Cysteine capsules based on number of drinks consumed and fill out a Hangover Symptom Scale the next morning
  Interventions: Dietary Supplement: N-acetyl cysteine

INTERVENTIONS:
Dietary Supplement: N-acetyl cysteine
  Arms: N-acetyl cysteine
Other: placebo
  Arms: Placebo

SUMMARY:
This is a double-blinded study involving healthy non-alcoholic (self-reported) volunteers over the age of 21. Consent is obtained prior to participation in the study while the participant is sober. Volunteers are recruited from residency programs, hospital employees, emergency medical personnel, and friends of the study investigators. If the volunteers choose to drink, they can participate in the study the night of ingestion of alcohol. There is no amount we ask them to drink, and we allow them to withdraw from the study at any time. We never force them to drink alcohol, or even encourage it. The participation is completely voluntary, if they would like to participate and if they choose to drink alcohol, we ask them to participate in the placebo controlled study in the safety of their own home. Then materials for the study are given out prior to their participation. An envelope is given with the questionnaire, and a small packet containing 3 pills of either NAC or placebo, and a small smear of Vicks vapor rub concealed in a small packet. At the end of their alcohol ingestion, the volunteer is asked to estimate the number roof drinks consumed and take 1 capsule per 3 drinks consumed of either 600 mg N-Acetyl-L-Cysteine or placebo capsules. In the morning, each participant fills out a Hangover Symptom Score questionnaire . A random number generator is used to determine placebo or NAC first, then the participant is given the other treatment at their subsequent encounter. Then study is being conducted over a series of many months, and data can be analyzed by the hangover symptoms scale data when using NAC compared to placebo. The data will be analyzed using the numerical values of each category for hangover classification and compare the placebo data to the control data.

ELIGIBILITY:
Inclusion Criteria:

* age over 21 years
* able and agrees to drink alcohol

Exclusion Criteria:

* alcoholism (self-reported)
* pregnancy
* reactive airway disease
* diabetes
* kidney/bladder stones
* kidney disease
* liver disease
* stomach ulcer
* organ transplant patients
* dialysis patients
* allergies to alcohol, eggs, milk, or wheat
* volunteers taking the following medications: opiate pain medication, activated charcoal, ampicillin,carbamazepine, cephalosporidine, methicillin, nitroglycerine, oxacillin, penicillin G, quinicillin

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Degree of hangover improvement as measured by hangover symptoms scale after using N-acetyl cysteine compared to placebo | less than 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's Hospital, Bethlehem, Pennsylvania, United States

REFERENCES:
- [Background] Lieber CS. Relationships between nutrition, alcohol use, and liver disease. Alcohol Res Health. 2003;27(3):220-31. PMID 15535450
- [Background] Swift R, Davidson D. Alcohol hangover: mechanisms and mediators. Alcohol Health Res World. 1998;22(1):54-60. PMID 15706734
- [Background] Gyamfi MA, Wan YJ. Pathogenesis of alcoholic liver disease: the role of nuclear receptors. Exp Biol Med (Maywood). 2010 May;235(5):547-60. doi: 10.1258/ebm.2009.009249. PMID 20463294